CLINICAL TRIAL: NCT04996667
Title: Study to Evaluate the Role of Inhaled Nitric Oxide (iNO) on Pulmonary Hemodynamics in Patients with Intermediate/submassive and Massive Pulmonary Embolism (PE)
Brief Title: Effect of INO in Patients with Submassive and Massive PE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no sponsor support
Sponsor: University of California, Los Angeles (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Principal Investigator, Rajan Saggar, Professor of Medicine, University of California, Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-000569
Record Dates: First submitted 2021-07-21; First posted 2021-08-09 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Pulmonary Embolism; Pulmonary Embolism Subacute Massive
MeSH Terms: conditions — Pulmonary Embolism | interventions — Endothelium-Dependent Relaxing Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Interventional Radiology Arm (Invasive Cohort) (Active Comparator): Interventional radiology (IR) will perform a right heart catheterization (RHC) as part of a planned IR procedure.
  Bedside apical 4 chamber view (RV:LV ratio) will be recorded using an ultrasound device, and noninvasive RV data will be obtained with Edwards ClearSight system and Edwards EV1000 clinical platform.
  The Butterfly iQ+ (one possible ultrasound device which may be used) is a single-probe, whole-body ultrasound device.
  After initial measurements, inhaled nitric oxide (iNO) will be administered at 30 ppm for 3 minutes. The same measurements will be obtained/calculated before, during iNO administration, and after iNO has been withheld for 2 minutes.
  Interventions: Drug: inhaled nitric oxide (iNO)
- Non-intervention Arm (Non-invasive Cohort) (Active Comparator): Vitals including O2 amount and modality, blood pressure, pressor name, dose, and rate will be recorded. If the patient is intubated, the name, dose, and rate of sedation and analgesia will be recorded. If the patient is not intubated, name and dose amount of sedation will be recorded. Arterial blood gas will be obtained if an A-line is placed. Bedside apical 4 chamber view will be recorded (RV:LV ratio) with an ultrasound device, and noninvasive RV data will be obtained with Edwards ClearSight system and Edwards EV1000 clinical platform. This data will be obtained before, during iNO administration, and after iNO has been withheld for 2 minutes.
  Interventions: Drug: inhaled nitric oxide (iNO)

INTERVENTIONS:
Drug: inhaled nitric oxide (iNO) — Inhaled nitric oxide (iNO), which is known mainly from the pulmonary hypertension literature for its therapeutic role in pulmonary arterial hypertension, has been proposed as a potential pharmacologic adjunct to standard anticoagulation in acute PE.
  Inhaled nitric oxide (iNO) will be administered at 30 ppm for 3 minutes. The measurements will be obtained/calculated before, during iNO administration, and after iNO has been withheld for 2 minutes.
  Other Names: INOmax

SUMMARY:
A single center study to evaluate the effect of inhaled nitric oxide (iNO) on pulmonary dynamics in patients presenting with imaging confirmed intermediate/submassive or massive pulmonary embolism (PE). The target enrollment is 20 subjects at Ronald Reagan UCLA Medical Center. PE patients undergoing catheter-based intervention will be administered iNO during their intervention and pulmonary hemodynamic measurement will be measured before, during, and after iNO administration (Invasive Cohort). Patients who are not undergoing catheter-based intervention will also be administered iNO and will have pulmonary hemodynamics, blood pressure, and heart rate measured non-invasively (Non-Invasive Cohort).

DETAILED DESCRIPTION:
This is a single center study to evaluate patients presenting with imaging confirmed intermediate/submassive or massive pulmonary embolism (PE). The investigators anticipate to enroll a total of 20-25 subjects at Ronald Reagan UCLA Medical Center.

After informed consent is obtained, the subject will proceed under one of two study intervention arms depending on his or her treatment plan. If the patient requires invasive treatment such as interventional thrombectomy or catheter-directed thrombolysis (CDT), the participant will be enrolled in the interventional radiology arm (invasive cohort). If the patient requires non-invasive treatment such as anticoagulation therapy, deep vein thrombosis (DVT) thrombectomy, or inferior vena cava (IVC) filter, the participant will be enrolled in the non-intervention arm (non-invasive cohort).

Interventional Radiology Arm (Invasive Cohort):

The following procedure will be performed:

Interventional radiology (IR) will perform a right heart catheterization (RHC) as part of a planned IR procedure. Patient arrives in the IR suite and is positioned flat with head of bed between flat and 45 degrees. O2 amount and modality, blood pressure, pressor name, dose, and rate will be recorded. If the patient is intubated, the sedation/analgesia drug name(s), dose(s), and rate(s) will be recorded. If the patient is not intubated, name and dose amount of sedation will be recorded. Arterial blood gas will be obtained if an A-line is placed.

Bedside apical 4 chamber view (RV:LV ratio) will be recorded using an ultrasound device, and noninvasive RV data will be obtained with Edwards ClearSight system and Edwards EV1000 clinical platform.

Edwards ClearSight system and Edwards EV1000 clinical platform is a finger probe worn with a supportive forearm strap. Hemodynamic measurements from the finger cuff will be recorded at intervals.

Novel non-invasive methods of estimating stroke volume and associated cardiac output have the potential to revolutionize PE risk stratification and care. Non-invasive blood pressure (NIBP) monitors can even measure stroke volume beat to beat, allowing for continuous evaluation of cardiac function. NIBP systems are typically composed of a finger cuff with an inflatable bladder, pressure sensors, and light sensors. An arterial pulse contour is formed using the volume clamp method of blood pressure measurement combined with calibration and brachial pressure reconstruction algorithms. The stroke volume with each heart beat can be estimated as the area under the systolic portion of the blood pressure curve divided by the afterload. A limitation of using NIBP monitors to measure stroke volume is their relative inaccuracy, as they are calculations of an indirect measurement. However, NIBP monitors¬ may improve clinical care of PE because they allow for assessment of dynamic cardiac changes in real time. Detection of worsening stroke volume in acute PE could inform providers of impending cardiac collapse, and improvement of stroke volume may function as a positive prognostic factor or marker of therapeutic success. Use of NIBP monitors during acute PE to identify clinically significant changes in cardiac function may advance both PE prognostication and management.

The Butterfly iQ+ (one possible ultrasound device which may be used) is a single-probe, whole-body ultrasound device.

After initial measurements, inhaled nitric oxide (iNO) will be administered at 30 ppm for 3 minutes. The same measurements will be obtained/calculated before, during iNO administration, and after iNO has been withheld for 2 minutes.

All major changes in pressures, sedation, vital signs, and major events will be recorded throughout the RHC procedure.

iNO is scheduled to be weaned off post RHC but the IR/anesthesia team may choose to keep the patient on iNO at their clinical discretion. The patient will then proceed to their standard of care IR procedures with planned intervention.

Non-intervention Arm (Non-invasive Cohort):

Vitals including O2 amount and modality, blood pressure, pressor name, dose, and rate will be recorded. If the patient is intubated, the name, dose, and rate of sedation and analgesia will be recorded. If the patient is not intubated, name and dose amount of sedation will be recorded. Arterial blood gas will be obtained if an A-line is placed. Bedside apical 4 chamber view will be recorded (RV:LV ratio) with an ultrasound device, and noninvasive RV data will be obtained with Edwards ClearSight system and Edwards EV1000 clinical platform. This data will be obtained before, during iNO administration, and after iNO has been withheld for 2 minutes.

If a subject initially enrolled in the Non-intervention Arm (Non-invasive Cohort) needs an invasive procedure, they will be removed from the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age.
* The patient or patient's surrogate decision maker must understand and sign the informed consent form (ICF).
* Hospitalized (Emergency Room (ER) or inpatient) with:
* Imaging (computed tomography pulmonary angiography (CTPA) or ventilation/perfusion (VQ) lung scan) proven acute pulmonary embolism (PE)
* PE meets the following intermediate risk PE criteria (or massive, see below):
* Troponin > .1 AND
* Imaging (computed tomography (CT) or transthoracic echocardiogram (TTE)) signs of RV compromise (at least 1 of the following):
* RV:LV>1 on TTE or CTPA OR RV dilation (TTE or CTPA OR RV dysfunction on TTE.
* Massive PE
* Intensive care unit (ICU) level of care (Patient moving to ICU, ICU level of care in ER, or currently in ICU)
* Ability to comply with study protocol in investigator's judgement

Exclusion Criteria:

* Pregnancy or breastfeeding
* Inability to administer iNO through current mode of O2 delivery (i.e. BiPAP)
* Active hemoptysis
* Known allergy to iNO.
* Any serious medical condition of lab abnormality that, in the investigator's judgement, precludes the patient's safe participation in the study.
* Methemoglobin reductase deficiency
* Unable to obtain consent or patient or patient surrogate decision maker declines
* Patients already on iNO prior to study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
right atrial pressure (RAP) | measured invasively during a right heart catheterization (RHC) before administration of iNO
  right atrial pressure (RAP) in mmHg
right atrial pressure (RAP) | measured invasively during a right heart catheterization (RHC) during administration of iNO
  right atrial pressure (RAP) in mmHg
right atrial pressure (RAP) | measured invasively during a right heart catheterization (RHC) after administration of iNO
  right atrial pressure (RAP) in mmHg
right ventricular pressure (RVP) | measured invasively during a right heart catheterization (RHC) before administration of iNO
  right ventricular pressure (RVP) in mmHg
right ventricular pressure (RVP) | measured invasively during a right heart catheterization (RHC) during administration of iNO
  right ventricular pressure (RVP) in mmHg
right ventricular pressure (RVP) | measured invasively during a right heart catheterization (RHC) after administration of iNO
  right ventricular pressure (RVP) in mmHg
pulmonary arterial pressure (PAP) | measured invasively during a right heart catheterization (RHC) before administration of iNO
  pulmonary arterial pressure (PAP) in mmHg
pulmonary arterial pressure (PAP) | measured invasively during a right heart catheterization (RHC) during administration of iNO
  pulmonary arterial pressure (PAP) in mmHg
pulmonary arterial pressure (PAP) | measured invasively during a right heart catheterization (RHC) after administration of iNO
  pulmonary arterial pressure (PAP) in mmHg
pulmonary capillary wedge pressure (PCWP) | measured invasively during a right heart catheterization (RHC) before administration of iNO
  pulmonary capillary wedge pressure (PCWP) in mmHg
pulmonary capillary wedge pressure (PCWP) | measured invasively during a right heart catheterization (RHC) during administration of iNO
  pulmonary capillary wedge pressure (PCWP) in mmHg
pulmonary capillary wedge pressure (PCWP) | measured invasively during a right heart catheterization (RHC) after administration of iNO
  pulmonary capillary wedge pressure (PCWP) in mmHg
cardiac output (CO) (by Fick and Thermodilution) | measured invasively during a right heart catheterization (RHC) before administration of iNO
  Cardiac Output (CO) is the amount of blood the heart pumps from each ventricle per minute. It is usually expressed in litres per minute (L/min).
cardiac output (CO) (by Fick and Thermodilution) | measured invasively during a right heart catheterization (RHC) during administration of iNO
  Cardiac Output (CO) is the amount of blood the heart pumps from each ventricle per minute. It is usually expressed in litres per minute (L/min).
cardiac output (CO) (by Fick and Thermodilution) | measured invasively during a right heart catheterization (RHC) after administration of iNO
  Cardiac Output (CO) is the amount of blood the heart pumps from each ventricle per minute. It is usually expressed in litres per minute (L/min).
cardiac index (CI) (by Fick and Thermodilution) | measured invasively during a right heart catheterization (RHC) before administration of iNO
  Cardiac index (CI) is the cardiac output proportional to the body surface area (BSA). The unit of measurement is litres per minute per square metre (L/min/m2).
cardiac index (CI) (by Fick and Thermodilution) | measured invasively during a right heart catheterization (RHC) during administration of iNO
  Cardiac index (CI) is the cardiac output proportional to the body surface area (BSA). The unit of measurement is litres per minute per square metre (L/min/m2).
cardiac index (CI) (by Fick and Thermodilution) | measured invasively during a right heart catheterization (RHC) after administration of iNO
  Cardiac index (CI) is the cardiac output proportional to the body surface area (BSA). The unit of measurement is litres per minute per square metre (L/min/m2).
mixed venous O2 | measured invasively during a right heart catheterization (RHC) before administration of iNO
  mixed venous O2 in %
mixed venous O2 | measured invasively during a right heart catheterization (RHC) during administration of iNO
  mixed venous O2 in %
mixed venous O2 | measured invasively during a right heart catheterization (RHC) after administration of iNO
  mixed venous O2 in %
central venous O2 | measured invasively during a right heart catheterization (RHC) before administration of iNO
  central venous O2 in %
central venous O2 | measured invasively during a right heart catheterization (RHC) during administration of iNO
  central venous O2 in %
central venous O2 | measured invasively during a right heart catheterization (RHC) after administration of iNO
  central venous O2 in %
systemic PaO2 | measured invasively during a right heart catheterization (RHC) before administration of iNO
  systemic PaO2 in mmHg
systemic PaO2 | measured invasively during a right heart catheterization (RHC) during administration of iNO
  systemic PaO2 in mmHg
systemic PaO2 | measured invasively during a right heart catheterization (RHC) after administration of iNO
  systemic PaO2 in mmHg
systolic blood pressure (SBP) | measured invasively during a right heart catheterization (RHC) before administration of iNO
  Systolic Blood Pressure in mmHg
systolic blood pressure (SBP) | measured invasively during a right heart catheterization (RHC) during administration of iNO
  Systolic Blood Pressure in mmHg
systolic blood pressure (SBP) | measured invasively during a right heart catheterization (RHC) after administration of iNO
  Systolic Blood Pressure in mmHg
diastolic blood pressure (DBP) | measured invasively during a right heart catheterization (RHC) before administration of iNO
  Diastolic Blood Pressure in mmHg
diastolic blood pressure (DBP) | measured invasively during a right heart catheterization (RHC) during administration of iNO
  Diastolic Blood Pressure in mmHg
diastolic blood pressure (DBP) | measured invasively during a right heart catheterization (RHC) after administration of iNO
  Diastolic Blood Pressure in mmHg
mean arterial pressure (MAP) | measured invasively during a right heart catheterization (RHC) before administration of iNO
  mean arterial pressure (MAP) in mmHg
mean arterial pressure (MAP) | measured invasively during a right heart catheterization (RHC) during administration of iNO
  mean arterial pressure (MAP) in mmHg
mean arterial pressure (MAP) | measured invasively during a right heart catheterization (RHC) after administration of iNO
  mean arterial pressure (MAP) in mmHg
blood pressure (BP) (measured noninvasively) | measured noninvasively before administration of inhaled nitric oxide (iNO)
  The pressure of the blood in the circulatory system, often measured for diagnosis since it is closely related to the force and rate of the heartbeat and the diameter and elasticity of the arterial walls.
  Systolic Blood Pressure in mmHg Diastolic Blood Pressure in mmHg
blood pressure (BP) (measured noninvasively) | measured noninvasively during administration of inhaled nitric oxide (iNO)
  The pressure of the blood in the circulatory system, often measured for diagnosis since it is closely related to the force and rate of the heartbeat and the diameter and elasticity of the arterial walls.
  Systolic Blood Pressure in mmHg Diastolic Blood Pressure in mmHg
blood pressure (BP) (measured noninvasively) | measured noninvasively after administration of inhaled nitric oxide (iNO)
  The pressure of the blood in the circulatory system, often measured for diagnosis since it is closely related to the force and rate of the heartbeat and the diameter and elasticity of the arterial walls.
  Systolic Blood Pressure in mmHg Diastolic Blood Pressure in mmHg
heart rate (HR) (measured noninvasively) | measured noninvasively before administration of inhaled nitric oxide (iNO)
  The number of heartbeats per unit of time, usually per minute.
  Measured in beats per minute (BPM)
heart rate (HR) (measured noninvasively) | measured noninvasively during administration of inhaled nitric oxide (iNO)
  The number of heartbeats per unit of time, usually per minute.
  Measured in beats per minute (BPM)
heart rate (HR) (measured noninvasively) | measured noninvasively after administration of inhaled nitric oxide (iNO)
  The number of heartbeats per unit of time, usually per minute.
  Measured in beats per minute (BPM)
cardiac index (CI) (measured noninvasively) | measured noninvasively before administration of inhaled nitric oxide (iNO)
  Cardiac index (CI) is the cardiac output proportional to the body surface area (BSA). The unit of measurement is litres per minute per square metre (L/min/m2).
cardiac index (CI) (measured noninvasively) | measured noninvasively during administration of inhaled nitric oxide (iNO)
  Cardiac index (CI) is the cardiac output proportional to the body surface area (BSA). The unit of measurement is litres per minute per square metre (L/min/m2).
cardiac index (CI) (measured noninvasively) | measured noninvasively after administration of inhaled nitric oxide (iNO)
  Cardiac index (CI) is the cardiac output proportional to the body surface area (BSA). The unit of measurement is litres per minute per square metre (L/min/m2).

CONTACTS AND LOCATIONS:
Overall Officials: Rajan Saggar, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- Ronald Reagan UCLA Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Summerfield DT, Desai H, Levitov A, Grooms DA, Marik PE. Inhaled nitric oxide as salvage therapy in massive pulmonary embolism: a case series. Respir Care. 2012 Mar;57(3):444-8. doi: 10.4187/respcare.01373. Epub 2011 Oct 12. PMID 22005573
- [Background] Capellier G, Jacques T, Balvay P, Blasco G, Belle E, Barale F. Inhaled nitric oxide in patients with pulmonary embolism. Intensive Care Med. 1997 Oct;23(10):1089-92. doi: 10.1007/s001340050461. PMID 9407246
- [Background] Szold O, Khoury W, Biderman P, Klausner JM, Halpern P, Weinbroum AA. Inhaled nitric oxide improves pulmonary functions following massive pulmonary embolism: a report of four patients and review of the literature. Lung. 2006 Jan-Feb;184(1):1-5. doi: 10.1007/s00408-005-2550-7. PMID 16598645
- [Background] Kline JA, Puskarich MA, Jones AE, Mastouri RA, Hall CL, Perkins A, Gundert EE, Lahm T. Inhaled nitric oxide to treat intermediate risk pulmonary embolism: A multicenter randomized controlled trial. Nitric Oxide. 2019 Mar 1;84:60-68. doi: 10.1016/j.niox.2019.01.006. Epub 2019 Jan 8. PMID 30633959